CLINICAL TRIAL: NCT05322850
Title: Phase I/II Trial: Engineered Donor Graft (Orca Q) for Pediatric Hematopoietic Cell Transplant (HCT) Recipients With Hematologic Malignancies (HM)
Brief Title: Phase I/II Trial: Engineered Donor Graft (Orca Q) for Pediatric Hematopoietic Cell Transplant (HCT)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Orca Biosystems, Inc. (Industry); Florida Department of Health (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UF-PED-003; OCR41968 (Other: University of Florida)
Record Dates: First submitted 2022-03-31; First posted 2022-04-12 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Acute Myeloid Leukemia; Acute Lymphoid Leukemia; Mixed Phenotype Acute Leukemia; Acute Undifferentiated Leukemia; Chronic Myeloid Leukemia in Myeloid Blast Crisis; Chronic Myeloid Leukemia in Lymphoid Blast Crisis (Diagnosis); Chronic Myeloid Leukemia - Accelerated Phase
Keywords: hematologic malignancies; Orca-Q; hematopoietic cell transplant; engineered donor graft; pediatrics
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Biphenotypic, Acute; Disease; Leukemia, Myeloid, Accelerated Phase; Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Orca-Q (Experimental)
  Interventions: Biological: Orca-Q

INTERVENTIONS:
Biological: Orca-Q — All transplant recipients enrolled on this study in both the phase I and phase II portions will receive Orca-Q (Orca-Q Prime and Orca-Q Supplement) intravenously following myeloablative conditioning.

SUMMARY:
This is a first in children prospective study of allogeneic hematopoietic cell transplant using a centrally manufactured engineered donor graft (Orca-Q). The study will assess safety and efficacy of Orca-Q in pediatric patients with hematologic malignancies.

ELIGIBILITY:
Inclusion Criteria (Recipients):

* Age < 22 years of age at the time of diagnosis of malignancy
* Eligible for treatment at a pediatric HCT center
* Patients with the following histopathologically-confirmed diseases are eligible:

  1. Acute myeloid, lymphoid, mixed phenotype or undifferentiated leukemia in complete remission (CR) or CR with incomplete hematologic recovery (CRi) as defined by:

     * Marrow blasts < 5% by morphologic examination
     * Absolute neutrophil count > 1.0 × 109/L
     * Platelet count > 100 × 109/L
     * Absence of leukemic blasts in the peripheral blood by morphological examination, and
     * No evidence of extramedullary disease
     * CRi: All CR criteria except for residual neutropenia (< 1.0 × 109/L) or thrombocytopenia (< 100 × 109/L)
  2. Myeloid or lymphoid blast crisis or accelerated phase developing in the setting of chronic myeloid leukemia is an allowed diagnosis provided that patients are in CR or CRi with regard to the blast crisis
* Planned to undergo myeloablative allogeneic hematopoetic cell transplant (MA-alloHCT) with a myeloablative conditioning regimen
* Available donor willing to donate PBSCs:

  1. Related donor who is a 7 or 8/8 match for HLA-A, -B, -C, and -DRB1, all typed using DNA-based high-resolution methods
  2. Matched unrelated donor who is a 7 or 8/8 match at HLA-A, -B, -C, and -DRB1, all typed using DNA-based high-resolution methods
  3. Haploidentical related donor who is a ≥ 4/8 but < 7/8 match at HLA-A, -B, -C, and -DRB1 (typed using DNA-based high-resolution methods), with at most one mismatch per locus
* Serum creatinine within normal range for age and estimated GFR by Schwartz equation >70 ml/min/1.73m2. If serum creatinine is higher than normal, obtain creatinine clearance or nuclear medicine glomerular filtration rate. GFR of ≥ 70 mL/minute/1.73m2 is required.
* Cardiac ejection fraction at rest ≥ 50% by echocardiogram or radionuclide scan (MUGA)
* Diffusing capacity of the lung for carbon monoxide (DLCO) (adjusted for hemoglobin) ≥ 70% or pulse ox on RA >95% for patients who cannot cooperate with the PFTs
* Total bilirubin < 1.5 times upper limit of normal (ULN) (< 3 times if attributed to Gilbert's syndrome) and ALT/AST < 4 times ULN
* Recipients in screening must screen negative for SARS-CoV-2 RNA using a PCR-based test prior to enrollment as follows:

  1. The SARS-CoV-2 testing screening test should be timed such that the results are available prior to the start of the recipient's conditioning regimen. Efforts should be made to minimize the window of time between test result availability and the start of conditioning.
  2. Recipients in screening who test positive for SARS-CoV-2 are ineligible but may be considered eligible for future trial participation provided that they are cleared for transplantation per the most current ASTCT guidelines (https://www.astct.org/connect/astct-response-to-covid-19).
* Subjects must not have more than one active malignancy at the time of enrollment (Subjects with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen [as determined by the treating physician and approved by the PI] may be included).
* Written informed consent obtained from the subject and the subject or parental/legal representative permission and subject's assent, if applicable, stating that the subject agrees to comply with all the study-related procedures.
* Women of childbearing potential (WOCBP) must be using an adequate method of contraception to avoid pregnancy throughout the study and for one year after transplantation to minimize the risk of pregnancy.
* Males with female partners of child-bearing potential must agree to use physician-approved contraceptive methods (e.g ., abstinence, condoms, vasectomy) throughout the study and should avoid conceiving children for one year after transplantation.

Inclusion Criteria (Donors):

* Age ≥ 18 and ≤ 50 years at time of enrollment
* Match to the patient as follows:

  1. Matched related donor who is a 7 or 8/8 match for HLA-A, -B, -C, and -DRB1, all typed using DNA-based high resolution methods
  2. Matched unrelated donor who is a 7 or 8/8 match at HLA-A, -B, -C, and -DRB1, all typed using DNA-based high-resolution methods
  3. Haploidentical related donor who is a ≥ 4/8 but < 7/8 match at HLA-A, -B, -C, and -DRB1 (typed using DNA-based high-resolution methods), with at most one mismatch per locus
* Willing to donate PBSC for up to two consecutive days
* Able to donate within North America or Hawaii at a site that will employ a Spectra Optia Apheresis System for post-mobilization apheresis.
* Meets federal eligibility criteria for donors of viable, leukocyte-rich cells or tissues as defined by 21 CFR § 1271 2018 and all relevant FDA Guidance for Industry.
* Donors determined to be ineligible, based on the results of required testing and/or screening, may nonetheless be included if either apply, as per 21 CFR § 1271.65 2018:

  1. The donor is a first-degree or second-degree blood relative of the recipient
  2. Urgent medical need, meaning no comparable human cell product is available and the Recipient is likely to suffer death or serious morbidity without the human cell product, as attested by the investigator.
* Meets any other criteria for donation as specified by standard NMDP guidelines (NMDP donors) or institutional/FACT standards (non-NMDP donors)

Exclusion Criteria (Recipients):

* Prior myeloablative allogeneic HCT
* Currently receiving corticosteroids or other immunosuppressive therapy (topical corticosteroids or physiologic replacement hydrocortisone is allowed)
* Planned donor lymphocyte infusion (DLI)
* Planned pharmaceutical in vivo or ex vivo T cell depletion, e.g., post-transplant cyclophosphamide (Cy) or alemtuzumab. Anti-thymocyte globulin is allowed only as specified in the protocol.
* Positive anti-donor HLA antibodies against a mismatched allele in the selected donor determined by either:

  1. a positive crossmatch test of any titer (by complement-dependent cytotoxicity or flow cytometric testing), or
  2. the presence of anti-donor HLA antibody to any of the following HLA loci: HLA-A, -B, -C, -DRB1, -DQB1, -DQA1, -DPB1, or -DPA1, with mean fluorescence intensity (MFI) > 1000 by solid phase immunoassay
* Lansky play scale < 70% or Karnofsky <70%
* Hematopoietic cell transplantation-specific Comorbidity Index (HCT-CI) > 4
* Documented or suspected bridging fibrosis or liver cirrhosis
* Uncontrolled bacterial, viral or fungal infections (currently taking antimicrobial therapy and with progression or no clinical improvement) at time of enrollment
* Seropositive for HIV-1 or -2, HTLV-1 or -2
* Known allergy or hypersensitivity to, or intolerance of, tacrolimus
* Documented allergy or hypersensitivity to iron dextran or bovine, murine, algal or Streptomyces avidinii proteins
* Any uncontrolled autoimmune disease requiring active immunosuppressive treatment
* Concurrent malignancies or active disease within 1 year, except non-melanoma skin cancers that have been curatively resected
* Females or males of childbearing potential who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period and for one year following transplantation.
* Females who are known to be pregnant or breastfeeding and unwilling to cease breastfeeding.
* Any serious medical condition or abnormality in clinical laboratory tests that, in the Investigator's or Medical Monitor's judgment, precludes the Recipient's safe participation in and completion of the study, or which could affect compliance with the protocol or interpretation of results
* Administration of a vaccine containing live virus within 30 days prior to the first dose of trial treatment (conditioning regimen). Note: Most flu vaccines are killed viruses, with the exception of the intra-nasal vainer (Flu-Mist) which is an attenuated live virus and therefore prohibited for 30 days prior to first dose. Non-live versions of the COVID-19 vaccine are allowed.
* Prisoners or subjects who are involuntarily incarcerated, wards of state, or subjects who are compulsorily detained for treatment of either a psychiatric or physical illness.

Exclusion Criteria (Donors):

* Evidence of active infection
* Seropositive for HIV -1 or -2, HTLV-1 or -2
* Positive for active or chronic Hepatitis B (HBV) based on serology [HBV surface antigen (HBsAg), total anti-Hepatitis B core antibody (HBcAb, IgG and IgM), and Hepatitis B surface antibody (HBsAb)] or by nucleic acid testing (NAT) testing. Donors with ambiguous HBV serology results should be tested for HBV by NAT.
* Positive for anti-Hepatitis C (HCV) antibody or HCV NAT
* Potential for Zika virus infection as defined as any of the following:

  * Medical diagnosis of Zika virus infection in the past 6 months
  * Residence in, or travel to, an area with active Zika virus transmission within the past 6 months.
  * Sex within the past 6 months with a person who is known to have either of the risk factors listed above
  * Donors determined to be ineligible based on the results of Zika virus screening may be determined to be eligible if:

    i. The donor has no signs or symptoms consistent with active Zika virus infection and either of the following is true: ii. The donor is a first-degree or second-degree blood relative of the recipient iii. Urgent medical need, meaning no comparable human cell product is available and the recipient is likely to suffer death or serious morbidity without the human cell product, as attested by the Investigator
* Aberrant CD45RA isoform expression by central laboratory testing
* Females who are pregnant or breastfeeding and unwilling to cease breastfeeding

Max Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-08-16 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Primary graft failure | 28 days
  Evaluate primary graft failure through day +28, defined as being alive without recovery of neutrophils (achieving an absolute neutrophil count >500/µL for 3 consecutive days) by day +28
Secondary graft failure | 100 days
  Evaluate secondary graft failure through day +100, defined as neutrophil engraftment followed by subsequent decline in absolute neutrophil counts to <500 µL, unresponsive to growth factor therapy and in the absence of alternative explanations such as recurrence of the underlying malignant disorder, infections, microangiopathy, medications causing bone marrow suppression or immune-mediated cytopenia.

SECONDARY OUTCOMES:
Non-relapse mortality (12 months post-transplant) | 12 months
  Evaluate non-relapse mortality, defined as death without evidence of disease recurrence, at 12 months post-transplant
Non-relapse mortality (24 months post-transplant) | 24 months
  Evaluate non-relapse mortality, defined as death without evidence of disease recurrence, at 24 months post-transplant.
Overall survival | 24 months
  Determine the overall survival at 24 months post-transplant, as defined as the time from the date of transplant to the date of death from any cause or, for surviving patients, to the date of last follow-up.
Relapse rate (12 months post-transplant) | 12 months
  Determine the relapse rate, as defined as the incidence of disease relapse through 12 months post-transplant. Disease relapse is defined as any of the following: ≥ 5% blasts in the bone marrow or peripheral blood, reappearance of pre-transplant cytogenetic abnormality, new evidence or redevelopment of extramedullary disease. Institution of any therapy to treat relapsed disease, such as withdrawal of immunosuppression or donor lymphocyte infusion (DLI), will be considered evidence of relapse regardless of whether any of these are met.
Relapse rate (24 months post-transplant) | 24 months
  Determine the relapse rate, as defined as the incidence of disease relapse through 24 months post-transplant. Disease relapse is defined as any of the following: ≥ 5% blasts in the bone marrow or peripheral blood, reappearance of pre-transplant cytogenetic abnormality, new evidence or redevelopment of extramedullary disease. Institution of any therapy to treat relapsed disease, such as withdrawal of immunosuppression or donor lymphocyte infusion (DLI), will be considered evidence of relapse regardless of whether any of these are met.
Rate of acute GVHD | 6 months
  Determine the rate of acute GVHD at 6 months post-transplant
Rate of chronic GVHD | 24 months
  Determine the rate of chronic GVHD through 24 months post-transplant.
Serious infection rate | 12 months
  Determine the rate of serious infections by 12 months post-transplant. A serious infection is defined as any new viral, bacterial, fungal or parasitic infection Common Terminology Criteria for Adverse Events v5.0 grade 2 or higher.
Treatment-Emergent Adverse Events | 24 months
  Describe treatment-emergent adverse events through 24 months post-transplant.
Graft-versus-host disease (GVHD)-free, relapse-free survival | 12 months
  Evaluate the GVHD-free, relapse-free survival at 12 months post-transplant. GVHD-free, relapse-free survival is defined as freedom from grade III or IV acute GVHD, moderate or severe chronic GVHD, or disease progression or relapse.

CONTACTS AND LOCATIONS:
Overall Officials: Jordan Milner, MD, Principal Investigator — University of Florida
Locations (4):
- United States (4):
  - University of Florida, Gainesville, Florida
  - University of Miami, Miami, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida